CLINICAL TRIAL: NCT02853110
Title: Hypofractionated Focal Lesion Ablative Microboost in prostatE Cancer (Hypo-FLAME)
Brief Title: Hypofractionated Focal Lesion Ablative Microboost in prostatE Cancer
Acronym: Hypo-FLAME
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: UMC Utrecht (Other)
Collaborators: The Netherlands Cancer Institute (Other); Universitaire Ziekenhuizen KU Leuven (Other); Radboud University Medical Center (Other)
Responsible Party: Principal Investigator, L.G.W. Kerkmeijer, MD, PhD, UMC Utrecht
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NL53719.041.15a
Record Dates: First submitted 2016-06-24; First posted 2016-08-02 (Estimated); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Prostate Cancer Adenocarcinoma
Keywords: MRI, stereotactic body radiotherapy, hypofractionation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypo-FLAME (Experimental): External beam radiotherapy, 5 additional MRI scans, blood sampling
  Interventions: Radiation: Hypo-FLAME study

INTERVENTIONS:
Radiation: Hypo-FLAME study — SBRT technique with 35 Gy in 5 weekly fractions and an additional simultaneously integrated focal boost to the tumor nodule(s) visible on MRI up to 50 Gy. In addition, patients will be asked to undergo 5 additional MRI scans (~15 min/scan) without contrast enhancement prior to each radiation session as well as blood sampling for translational research (radiogenomics) and Biobank purposes.

SUMMARY:
The hypo-FLAME study is a multicenter phase II study (n=100) to investigate whether a focal SBRT boost to the MRI-defined macroscopic tumor volume is feasible and associated with acceptable toxicity in addition to whole gland prostate SBRT.

DETAILED DESCRIPTION:
Rationale: Hypofractionation with a stereotactic body radiotherapy (SBRT) technique for prostate cancer produces excellent treatment outcome in terms of survival and toxicity and is much more convenient than the current fractionation scheme. Local recurrence occurs most frequently at the site of the primary or dominant tumor location prior to treatment. Therefore dose escalation at the site of the primary tumor may improve disease control.

Objective: The main goal of this phase II study is to investigate whether a focal ablative SBRT boost to the macroscopic tumor is feasible and associated with acceptable toxicity in addition to whole gland prostate SBRT. The secondary objectives of this study are: late toxicity, quality of life (QoL) and biochemical disease free survival (bDFS). Furthermore, two side-studies are incorporated in this phase II study: 1) a weekly MRI will be performed to prepare for future MRI-guided (MR-linac) treatment without gold fiducial markers and 2) blood sampling for translational research (radiogenomics) and Biobank purposes.

Study design: Prospective multicenter interventional study on whole gland prostate SBRT using MRI for focal boost in 100 consecutive intermediate or high risk prostate cancer patients.

Study population: One hundred patients with histologically proven prostate adenocarcinoma with intermediate risk or high risk disease. Patients referred for external beam radiotherapy (EBRT) who fulfill the inclusion criteria and without any of the exclusion criteria will be included in the present trial after written informed consent.

Intervention: Patients will be treated by external beam radiotherapy with a SBRT technique with 35 Gy in 5 weekly fractions and an additional simultaneously integrated focal boost to the tumor nodule(s) visible on MRI up to 50 Gy. In addition, patients will be asked to undergo 5 additional MRI scans (~15 min/scan) without contrast enhancement prior to each radiation session as well as blood sampling for translational research (radiogenomics) and Biobank purposes.

Main study parameters/endpoints: The primary endpoints of this study are acute gastrointestinal (GI) and genitourinary (GU) toxicity using the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Secondary endpoints are late GI and GU toxicity, QoL, and bDFS. Simultaneously, two side-studies will be performed, i.e. to prepare for MRI-guided radiotherapy and blood sampling for translational research (radiogenomics) and Biobank purposes.

ELIGIBILITY:
Inclusion Criteria:

* Men ≥ 18 years with histologically confirmed prostate adenocarcinoma
* Intermediate-risk prostate cancer or high-risk prostate cancer, defined as at least one of the following risk criteria: clinical T-stage T2b, T2c or T3a (defined on MRI) or T3b with less than 5 mm invasion in the seminal vesicle, Gleason sum score ≥ 7, PSA ≥ 10 ng/mL
* Prostate tumor nodule visible on MRI
* Ability to give written informed consent and willingness to return for follow-up

Exclusion Criteria:

* Prior pelvic radiotherapy, transurethral prostate resection or prostatectomy
* Unsafe to have gold fiducial marker implantation
* Contraindications to MRI according to the Radiology Department guidelines (metal implants, non-compatible cardiac device, allergy to Gadolinium, severe renal dysfunction or severe claustrophobia)
* Evidence of lymph node involvement or distant metastatic disease
* Clinical T-stage > T3b with ≥ 5 mm invasion in the seminal vesicle
* World Health Organization (WHO) performance score > 2
* International prostate symptoms score (IPSS score) ≥ 15
* PSA > 30 ng/mL

Ages: 18 Years to 100 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Acute toxicity | 90 days after first radiation treatment
  The goal of the present study is to investigate whether a focal SBRT boost to the macroscopic tumor is feasible and associated with acceptable toxicity in addition to whole gland prostate SBRT. Toxicity will be assessed by the acute gastrointestinal (GI) and genitourinary (GU) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Acute toxicity is defined as toxicity occurring within 90 days after the first radiation treatment.

SECONDARY OUTCOMES:
Late toxicity | 10 years after last radiation treatment
  Late toxicity, assessed by the late GI and GU Common Terminology Criteria for Adverse Events (CTCAE) version 4.0. Late toxicity is defined as toxicity occurring after at least 90 days after the first radiation treatment.
Quality of life - general | 5 years after last radiation treatment
  European Organisation for Research and Treatment of Cancer (EORTC) QLQ-C30 questionnaire
Biochemical disease free survival (bDFS) | 10 years after last radiation treatment
  Biochemical disease free survival
Quality of life - prostate specific | 5 years after last radiation treatment
  EORTC QLQ- PR25 questionnaire

OTHER OUTCOMES:
MRI side study | Within 5 weeks from start of radiotherapy
  Quantify intrafraction motion of the prostate (in mm)
Blood sampling | Within 5 weeks from start of radiotherapy
  Radiogenomic analyses

CONTACTS AND LOCATIONS:
Overall Officials: Linda GW Kerkmeijer, MD, PhD, Principal Investigator — UMC Utrecht
Locations (4):
- UZ Leuven, Leuven, Belgium
- Netherlands (3):
  - NKI-AvL, Amsterdam
  - Radboudumc, Nijmegen
  - UMC Utrecht, Utrecht

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Goodman CD, Fakir H, Pautler S, Chin J, Bauman GS. Dosimetric Evaluation of PSMA PET-Delineated Dominant Intraprostatic Lesion Simultaneous Infield Boosts. Adv Radiat Oncol. 2019 Sep 27;5(2):212-220. doi: 10.1016/j.adro.2019.09.004. eCollection 2020 Mar-Apr. PMID 32280821
- [Derived] Draulans C, van der Heide UA, Haustermans K, Pos FJ, van der Voort van Zyp J, De Boer H, Groen VH, Monninkhof EM, Smeenk RJ, Kunze-Busch M, De Roover R, Depuydt T, Isebaert S, Kerkmeijer LGW. Primary endpoint analysis of the multicentre phase II hypo-FLAME trial for intermediate and high risk prostate cancer. Radiother Oncol. 2020 Jun;147:92-98. doi: 10.1016/j.radonc.2020.03.015. Epub 2020 Apr 1. PMID 32247206